CLINICAL TRIAL: NCT04285138
Title: Effects of Phantom Exercises on Pain, Mobility and Quality of Life Among Lower Limb Amputees
Brief Title: Phantom Exercise for Lower Limb Amputees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/20/2008 Anna Zaheer
Record Dates: First submitted 2020-02-24; First posted 2020-02-26 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Lower Limb Amputation
Keywords: Phantom; Amputation; Prosthesis

STUDY DESIGN:
Intervention Model Description: Phantom exercises involved imagining moving the phantom limb and then attempting to perform these movements
  The phantom exercises will be administered as follows:
  (i) subjects will be asked in which position they felt the phantom limb; (ii) they will be asked to place the intact limb in the same position as they felt their phantom limb; (iii) they will be asked to move both limbs in the opposite direction; (iv) they will be then asked to return to the starting position again.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phantom limb exercises (Experimental): Participants in this group will be treated with routine physical therapy, mirror therapy and Phantom limb exercises. Treatment time: 1 hour
  Interventions: Other: phantom limb exercise
- conventional treatment (Active Comparator): In this group, participants will be treated by routine physical therapy and mirror therapy protocol. Treatment time: 35 minutes
  Interventions: Other: conventional treatment

INTERVENTIONS:
Other: phantom limb exercise — phantom limb exercises (that is, active imaginal efforts to move the phantom), under the assumption that the neural pathways involved in performing actual movements are activated when using one's imagination to move the phantom extremity
  Arms: Phantom limb exercises
Other: conventional treatment — Mirror therapy uses a flat mirror placed parasagittally in front of the patient's body with the reflective surface toward the sound limb so that the amputee sees the reflection of the sound limb in the mirror [Figure 1]. This reflection mimics the amputated limb, and with the movement of the intact limb, the mirror provides an optical illusion that the phantom limb is moving simultaneously.
  Equipment:
  Therapy mirror: A standing mirror (130 cm × 46 cm) with wooden frame and base (62 cm × 65 cm) Routine physiotherapy The general exercise programme consisted of strengthening, stretching, dynamic, and isometric exercises based on the level of amputation and their assessment results. Participants allocated to the control group were advised to continue rehabilitation at their respective physiotherapy out-patient departments as frequently as possible. Participants were given a diary and advised to record their activities, specifying the nature, frequency and duration of each activity
  Arms: conventional treatment

SUMMARY:
In this research, the aim is to find out the effects of phantom exercises in terms of pain, mobility and quality of life among lower-limb amputees having phantom limb pain. This is a randomized control trial in which amputees having phantom limb pain will be randomly divided into two groups i.e. Experimental group (Routine physical therapy, mirror therapy and phantom exercises) and control group (Routine physical therapy and mirror therapy). Non-probability purposive sampling technique will be employed. Patients of age between 18 to 50 years and having phantom limb pain after lower limb amputation will be recruited by evaluating with limb deficiency and phantom limb questionnaire. Other tools will be Visual analogue scale (pain), Amputee mobility predictor (Ambulatory status) and 36-Item Short-Form Health Survey questionnaire (Health-related quality of life). The study will be conducted in 6 months and data obtained will be analyzed through Statistical Package for Social Sciences (SPSS) 20.

DETAILED DESCRIPTION:
An amputation is a distressing event that will result in physical, psychological, and social consequences. The loss of limb means a huge impact, not only for the patient's body and the way he notices it, as well as the perception of the environment around him. Most of the patients with lower extremity amputations experienced phantom limb pain. It is defined by painful sensation in the missing limb. According to a recent study, the prevalence of phantom limb pain ranges from 45% to 85%. Regardless of the reason for amputation, phantom limb pain diminishes over time in most cases. However, in about 5-10% of amputees' severe pain persists for several years. It affects the patient's capacity for self-care and personal independence as it is mentally and physically debilitating. Incidence of PLP in recent studies is reported to be approximately 42.2-78.8% of amputees. It should be noted that phantom limb pain (PLP) differs from pain in the stump called residual limb pain (RLP), which is due to skin complications, vascular compromise, inappropriate healing, painful neuromas, excess soft tissue and bone irregularities.

However, the exact mechanism of phantom limb pain is unknown, but advancement in pain physiology indicates that multiple mechanisms are involved including peripheral, spinal and supraspinal mechanisms. The first changes may take place in the periphery where the nerve endings are sensitized by pre-amputation pain and nerve transection. But the complexity of phantom phenomena and the association between catastrophizing and phantom limb pain indicate that supraspinal changes play a significant role in phantom pain. It is likely that the relative contributions of these mechanisms vary from one amputee to another and that they may change over time in the individual patient.

It has been seen that phantom limb pain is typically experienced in regions with large cortical representation, such as the hands/fingers and feet/toes. The pain is often described with words such as knifelike, sticking, pricking, shooting, and burning. Both PLP and RLP have a high incidence among amputees. These pains are a continual reminder of circumstances and can affect important factors of Quality of life such as sleep, fatigue mood and relationships compromising the acquisition of skills and quality of life. Thus, interfering with the physical and psychosocial rehabilitation of the amputee. This should be considered clinically during therapeutic encounters, and amputees should be given appropriate information on these potential associations, though often neglected by the medical team. Although QOL in amputees seems primarily determined by mobility impairment, pain, emotional perturbation, it is seen that physician-controlled factors such as the timing of amputation, informed decision making, and postamputation support may also play an important role. This data can be efficiently collected through limb deficiency and phantom limb questionnaire. During the rehabilitation process, multiple tools are available that help physicians to determine both motor ability and mobility in amputees as well as other determinants of quality of life and pain status of amputees. These include tests that determine motor ability as Single-limb standing balance test (Balance test), the Lower-Extremity Motor Coordination Test (LEMOCOT) and the Amputee Mobility Predictor without a prosthesis (AMPnoPRO). The AMP is a highly reliable instrument and it is relatively easy to administer in 15 minutes or less. Patients characteristics can be easily evaluated using "Limb Deficiency and Phantom Limb Questionnaire (Questionnaire 2008, Version 2)" and visual analogue scale (VAS) for the presence and extent of PLP. Health-related quality of life (HRQL) will be measured by the SF-36 questionnaire.

Despite a growing body of evidence, phantom limb pain remains a challenging condition to treat. There remains a large potential for innovation in improving the treatment strategies for these patients. More than 25 treatments for PLP are currently available yet not one is widely accepted or superior to others. Common self-treatment strategies can include wearing an elastic stump sock to minimise volume changes in the residual limb, stump massage, mental imagery of the phantom limb and taking physical exercise.

A rehabilitation technique that proved promising in recent years is mirror therapy, which involves a mirror being placed in a position that allows the patient to view a reflection of a body part. whilst the nonpainful limb is placed in front of the mirror so that it creates a reflection that can be seen by the patient, the stump is kept behind the mirror. In amputees, this creates the illusion of having two intact limbs and then the patient is asked to move an intact limb in certain patterns. This gives the illusion that the painful limb can move normally too. The mechanism of action of mirror therapy remains uncertain, with the reintegration of motor and sensory systems, restored body image and control over fear-avoidance likely to influence the outcome. Nevertheless, mirror therapy is inexpensive, safe and easy for the patient to self-administer but the level of evidence is insufficient. A limitation of the mirror box technique is the poor verisimilitude of the sensory feedback provided from the missing limb. The participant may have the visual illusion that the phantom extremity is moving, but the apparatus is crude and the illusion often not compelling. Patients cannot independently control the mirrored extremity, so only symmetric actions can be modelled.

Moreover, a relatively less researched method of reduction of phantom limb pain is Phantom exercises (PE). This involved imagining moving the phantom limb and then attempting to perform a few movements. The neurophysiological network activated during phantom limb movements is similar to that of executed movements of intact limbs and differs from the phantom limb imagination network. The dual ability of amputees to execute and imagine movements of their phantom limb and the fact that these two tasks activate distinct cortical networks are important factors to consider when designing rehabilitation programmes for the treatment of phantom limb pain. Few studies indicate that phantom exercises can be used safely to alleviate phantom limb pain in lower and upper limb amputees.

The evidence for clinical efficacy of mirror therapy is encouraging, but not yet definitive. Virtual reality could be a substitute for mirror therapy especially in the case if person suffers from bilateral amputation but even though the use of an immersive virtual reality (VR) environment may have a short-term effect on PLP for the majority of amputees who experience PLP, it's cost remain a problem in developing country like Pakistan, Moreover, because of high prevalence and high pain intensity of phantom limb pain, there is need to find an effective, easily administered home-based treatment for amputees, thus comparing effects of mirror therapy with and without phantom exercises in reducing pain and improving QOL and psychological status of amputees is a useful guide for future studies as these protocols are cost-effective and efficient.

In a pilot, study authors investigated the effects of phantom limb exercises on phantom limb pain. A total of 20 traumatic amputees participated in the study. Ten received phantom exercises and prosthetic training, and 10 were treated with routine prosthetic training and a general exercise programme. They found that pain intensity decreased in all subjects after 4 weeks of treatment in both groups. according to the visual analogue scale scores at the end of 4 weeks, the phantom exercises group differed significantly from the general exercise group. Thus, the study indicated that phantom exercises can be used safely to alleviate phantom limb pain in lower and upper limb amputees.

This study combines the effect of mirror therapy with phantom exercises in the experimental group. Similarly, another randomized controlled trial (RCT) was done to evaluate the reduction in phantom pain and sensation with combined training of progressive muscle relaxation, mental imagery and phantom exercises. This randomized controlled prospective trial with two parallel groups included Fifty-one subjects with unilateral lower limb amputation with Phantom Limb Pain. The experimental group performed combined training of progressive muscle relaxation, mental imagery and phantom exercises 2 times a week for 4 weeks, while the control group had the same amount of physical therapy dedicated to the residual limb. The results showed a significant decrement over time in all the Patient evaluation questionnaire domains (both in terms of phantom limb sensation (PLS) and phantom limb pain (PLP) and Brief pain intensity in experimental groups. The conclusion of this suggested that combined training of progressive muscle relaxation, mental imagery and modified phantom exercises should be taken into account as a valuable technique to reduce phantom limb pain and sensation. As Mirror therapy (MT) has been proposed as an effective rehabilitative strategy to alleviate pain symptoms in amputees with phantom limb pain (PLP) so in this study mirror therapy is used as conventional treatment along with the general exercise programme for amputees.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral lower limb amputation
* Phantom limb pain score (40-100 on VAS)
* Either gender
* Stable prosthetic situation (i.e. satisfaction with the fitting of the prosthesis) or being a non-user.

Exclusion Criteria:

* Amputees with psychological/neurological impairments.
* Amputees having neuropathic pain other than phantom limb pain.
* Patients having visual-spatial impairments.
* Taking pain relief medications will also be excluded.
* Patients having residual limb pain.
* Inability to give informed consent.
* Carcinoma
* Infectious stump
* Severe hearing loss
* Any condition that restricts the movement of opposite limb, pain or limited range of motion in the intact limb
* Infectious and systematic diseases

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) | 4 weeks
  changes from the baseline, The visual analogue scale The VAS evaluates pain subjectively. It consists of a 100-mm line, with two endpoints representing "no pain" to "worst pain imaginable from left to right." Patients are instructed to mark on the line according to the level of pain and the same is measured
Amputee Mobility predictor | 4 weeks
  changes from the baseline, Amputee mobility predictor (AMP) is an amputee-specific tool for predicting ambulatory potential. This clinical test evaluates the predicted mobility of amputee with and without a prosthesis The AMP is a clinical test consisting of 20 tasks that are given a score of 0, 1, or 2 based on the amputee's performance. There is an item 21 where a score is given ranging from 0 to 5.
Limb Deficiency and Phantom Limb Questionnaire | day 1
  Patients will be evaluated using "Limb Deficiency and Phantom Limb Questionnaire (Questionnaire 2008, Version 2)" in order to assess their eligibility for including in this study.
  this questionnaire does not have any scoring, it only concludes the questions on Yes/No basis for presence or absence of phantom limb pain.

SECONDARY OUTCOMES:
Short form 36 (SF-36) | 4 weeks
  changes from the baseline, The 36-Item Short-Form Health Survey questionnaire (SF-36) is a very popular instrument for evaluating Health-Related Quality of life (HRQOL). It is a widely used valid and reliable tool for measuring the (HRQOL) and it can be employed in both the healthy and diseased population such as amputees for assessing the outcome of health care services and the effect of medical intervention.
  The SF-36 measures eight scales: physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MH). Component analyses showed that there are two distinct concepts measured by the SF-36: a physical dimension, represented by the Physical Component Summary (PCS), and a mental dimension, represented by the Mental Component Summary (MCS).

CONTACTS AND LOCATIONS:
Overall Officials: Arshad Nawaz Malik, PhD, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Solarz MK, Thoder JJ, Rehman S. Management of Major Traumatic Upper Extremity Amputations. Orthop Clin North Am. 2016 Jan;47(1):127-36. doi: 10.1016/j.ocl.2015.08.013. PMID 26614927
- [Background] Kuffler DP. Coping with Phantom Limb Pain. Mol Neurobiol. 2018 Jan;55(1):70-84. doi: 10.1007/s12035-017-0718-9. PMID 28921418
- [Background] Ayoub SN, Hakim KY. Comparative study of dexmedetomidine or fentanyl as an adjuvant to epidural bupivacaine for prevention of stump and phantom pain in adult patients undergoing above-knee or below-knee amputation: a randomized prospective trial. Research and Opinion in Anesthesia and Intensive Care. 2019;6(3):371
- [Background] Padovani MT, Martins MR, Venancio A, Forni JE. Anxiety, depression and quality of life in individuals with phantom limb pain. Acta Ortop Bras. 2015 Mar-Apr;23(2):107-10. doi: 10.1590/1413-78522015230200990. PMID 27069411
- [Background] Nikolajsen L, Christensen KF. Phantom limb pain. Nerves and Nerve Injuries: Elsevier; 2015. p. 23-34.
- [Background] Hall N, Abd-Elsayed A, Eldabe S. Phantom Limb Pain. Pain: Springer; 2019. p. 907-10.
- [Background] Roberts K. The Role of Positivity: Physical and Mental Aspects of Lower Limb Amputation Due to Diabetes. 2019
- [Background] Trevelyan EG, Turner WA, Robinson N. Perceptions of phantom limb pain in lower limb amputees and its effect on quality of life: a qualitative study. Br J Pain. 2016 May;10(2):70-7. doi: 10.1177/2049463715590884. Epub 2015 Jun 23. PMID 27551416
- [Background] Suckow BD, Goodney PP, Nolan BW, Veeraswamy RK, Gallagher P, Cronenwett JL, Kraiss LW. Domains that Determine Quality of Life in Vascular Amputees. Ann Vasc Surg. 2015;29(4):722-30. doi: 10.1016/j.avsg.2014.12.005. Epub 2015 Feb 26. PMID 25725279
- [Background] Gailey RS, Roach KE, Applegate EB, Cho B, Cunniffe B, Licht S, Maguire M, Nash MS. The amputee mobility predictor: an instrument to assess determinants of the lower-limb amputee's ability to ambulate. Arch Phys Med Rehabil. 2002 May;83(5):613-27. doi: 10.1053/apmr.2002.32309. PMID 11994800
- [Background] Ramadugu S, Nagabushnam SC, Katuwal N, Chatterjee K. Intervention for phantom limb pain: A randomized single crossover study of mirror therapy. Indian J Psychiatry. 2017 Oct-Dec;59(4):457-464. doi: 10.4103/psychiatry.IndianJPsychiatry_259_16. PMID 29497188
- [Background] Pereira ÂM, Ramos A, Rafaela A, João M, Arrifes V. Mobility in patients with lower limb amputation after prosthesis. Annals of Medicine. 2019;51(sup1):212-.
- [Background] Aternali A, Katz J. Recent advances in understanding and managing phantom limb pain. F1000Res. 2019 Jul 23;8:F1000 Faculty Rev-1167. doi: 10.12688/f1000research.19355.1. eCollection 2019. PMID 31354940
- [Background] Le Feuvre P, Aldington D. Know pain know gain: proposing a treatment approach for phantom limb pain. J R Army Med Corps. 2014 Mar;160(1):16-21. doi: 10.1136/jramc-2013-000141. Epub 2013 Jul 31. PMID 24109117
- [Background] Wittkopf PG, Johnson MI. Mirror therapy: A potential intervention for pain management. Rev Assoc Med Bras (1992). 2017 Nov;63(11):1000-1005. doi: 10.1590/1806-9282.63.11.1000. PMID 29451665
- [Background] Barbin J, Seetha V, Casillas JM, Paysant J, Perennou D. The effects of mirror therapy on pain and motor control of phantom limb in amputees: A systematic review. Ann Phys Rehabil Med. 2016 Sep;59(4):270-5. doi: 10.1016/j.rehab.2016.04.001. Epub 2016 May 30. PMID 27256539
- [Background] Ambron E, Miller A, Kuchenbecker KJ, Buxbaum LJ, Coslett HB. Immersive Low-Cost Virtual Reality Treatment for Phantom Limb Pain: Evidence from Two Cases. Front Neurol. 2018 Feb 19;9:67. doi: 10.3389/fneur.2018.00067. eCollection 2018. PMID 29515513
- [Background] Raffin E, Mattout J, Reilly KT, Giraux P. Disentangling motor execution from motor imagery with the phantom limb. Brain. 2012 Feb;135(Pt 2):582-95. doi: 10.1093/brain/awr337. PMID 22345089
- [Background] Ulger O, Topuz S, Bayramlar K, Sener G, Erbahceci F. Effectiveness of phantom exercises for phantom limb pain: a pilot study. J Rehabil Med. 2009 Jun;41(7):582-4. doi: 10.2340/16501977-0380. PMID 19543671
- [Background] Brunelli S, Morone G, Iosa M, Ciotti C, De Giorgi R, Foti C, Traballesi M. Efficacy of progressive muscle relaxation, mental imagery, and phantom exercise training on phantom limb: a randomized controlled trial. Arch Phys Med Rehabil. 2015 Feb;96(2):181-7. doi: 10.1016/j.apmr.2014.09.035. Epub 2014 Oct 23. PMID 25450123
- [Background] Saleh Velez FG, Pinto CB, Bailin ES, Munger M, Ellison A, Costa BT, Crandell D, Bolognini N, Merabet LB, Fregni F. Real-time Video Projection in an MRI for Characterization of Neural Correlates Associated with Mirror Therapy for Phantom Limb Pain. J Vis Exp. 2019 Apr 20;(146):10.3791/58800. doi: 10.3791/58800. PMID 31058883
- [Background] Pandian JD, Rajni Arora M, Kaur P. Mechanisms underlying mirror therapy and its clinical applications. 2019.
- [Background] Anaforoglu Kulunkoglu B, Erbahceci F, Alkan A. A comparison of the effects of mirror therapy and phantom exercises on phantom limb pain. Turk J Med Sci. 2019 Feb 11;49(1):101-109. doi: 10.3906/sag-1712-166. PMID 30762318
- [Background] Davie-Smith F, Paul L, Stuart W, Kennon B, Young R, Wyke S. The Influence of Socio-economic Deprivation on Mobility, Participation, and Quality of Life Following Major Lower Extremity Amputation in the West of Scotland. Eur J Vasc Endovasc Surg. 2019 Apr;57(4):554-560. doi: 10.1016/j.ejvs.2018.10.011. Epub 2019 Mar 21. PMID 30905506
- [Background] Yaqoob I, Khalil K, Fayyaz R, Khan A. Functional ability and quality of life of below knee amputees with prosthesis. Rawal Medical Journal. 2018;43(4):708-11.
- [Background] Alghadir AH, Anwer S, Iqbal A, Iqbal ZA. Test-retest reliability, validity, and minimum detectable change of visual analog, numerical rating, and verbal rating scales for measurement of osteoarthritic knee pain. J Pain Res. 2018 Apr 26;11:851-856. doi: 10.2147/JPR.S158847. eCollection 2018. PMID 29731662
- [Derived] Zaheer A, Malik AN, Masood T, Fatima S. Effects of phantom exercises on pain, mobility, and quality of life among lower limb amputees; a randomized controlled trial. BMC Neurol. 2021 Oct 27;21(1):416. doi: 10.1186/s12883-021-02441-z. PMID 34706654